CLINICAL TRIAL: NCT02812446
Title: Staphylokinase and ABO Group Phenotype: New Players in Staphylococcus Aureus Implant-associated Infections Development
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC15_0456
Record Dates: First submitted 2016-06-16; First posted 2016-06-24 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Staphylococcal Infection
Keywords: biofilm; staphylokinase; Staphylococcus aureus; microarrays; bone binding sialoprotein; bone and joint infection; blood group
MeSH Terms: conditions — Staphylococcal Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — A total of 57 nonduplicate S. aureus clinical isolates collected from implant-associated infections (IAI) between January 2007 and December 2010 at Nantes University Hospital (France) were analyzed. IAI were confirmed using Infectious Diseases Society of America criteria for bone and joint infections. Thirty-five isolates came from hip arthroplasty, 18 from knee replacement and four from osteosynthesis. Thirty-one S. aureus isolates were collected from 100 noninfected patients screened for S. aureus nasal colonization from December 2011 to February 2012 at the orthopedic consultation ward.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- IAI patients group: patients with Staphylococcus aureus of implant-associated infections
  Interventions: Other: IAI infection
- control group: patients with Staphylococcus aureus nasal carriage
  Interventions: Other: Staphylococcus aureus nasal carriage infection

INTERVENTIONS:
Other: IAI infection
  Groups: IAI patients group
Other: Staphylococcus aureus nasal carriage infection
  Groups: control group

SUMMARY:
The purpose of this study is to identify bacterial and/or clinical features involved in the pathogenesis of Staphylococcus aureus implant-associated infections (IAI). Materials & methods: In total, 57 IAI S. aureus and 31 nasal carriage (NC) S. aureus isolates were studied. Staphylococcus aureus genetic background was obtained by microarray analysis. Multilocus sequence typing was performed to determine clonal complexes (CC). Biofilm production was investigated by resazurin and crystal violet methods

ELIGIBILITY:
Inclusion Criteria:

* infected patients with S. Aureus IAI infection
* noninfected patients screened for S. aureus nasal colonization at the orthopedic consultation ward

Exclusion Criteria:

* minor

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Fifty-five IAI patients were included; two of them had two different S. aureus IAI episodes. The median age was 73 years (range: 21-96 years) with 29 women (52.7%). Twenty seven percent of patients suffered from diabetes and were smokers.
  Nine patients including six women were immunosuppressed with a median age of 71 years. The main diagnosis for arthroplasty was arthrosis (38%). Implants were hip prosthesis (n = 35), knee prosthesis (n = 18) and osteosynthesis (n = 4). Main local consequences of IAI were scarce alteration (n = 34) and skin fistulization (n = 22). These IAI were treated by surgical removal of all infected tissue and implant or a combination of debridement with implant retention associated to long-term antimicrobial therapy active against biofilm microorganisms. Eighteen early, nine delayed and 30 late infections occurred. Blood group phenotypes were available for 54 patients and were distributed as follows: 26 O group, 17 A group, 10 B group and one AB group.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2012-02; Primary Completion 2012-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
biofilm production measurement in the two groups | september 2012
  The primary aim of this study is to identify phenotypic (biofilm production) markers in two different groups of S. aureus strains isolated from patients with IAI or screened from nasal carrier in noninfected patients undergoing orthopedic surgery.
  By using resazurin method, IAI and NC nasal carriage isolates were divided into three groups. Isolates were classified as strong, moderate and weak biofilm producers.
Clonal complexes distribution | september 2012
  The primary aim of this study is to identify genotypic markers in two different groups of S. aureus strains isolated from patients with IAI or screened from nasal carrier in noninfected patients undergoing orthopedic surgery.
  IAI and NC isolates genetic background was determined in order to compare the prevalence of individual virulence factor genes. All genes provided by the Alere StaphyType DNA microarray were studied.
IAI and NC nasal carriage isolates genetic background | september 2012
  IAI and NC isolates genetic background was determined in order to compare the prevalence of individual virulence factor genes. All genes provided by the Alere StaphyType DNA microarray were studied

SECONDARY OUTCOMES:
biofilm production correlation with genotype | december 2013
  quantile-quantile (QQ)-plot analysis
Correlation between Clonal Complexes distribution , genotype and clinical parameters | december 2013
  In order to determine whether clusters of S. aureus could be associated with clinical characteristics of the patients, search of association between CCs and clinical data was performed
Association of ABO group phenotype and IAI S. aureus genotype | december 2013
  QQ-plots analysis

IPD SHARING:
Plan to Share IPD: No